CLINICAL TRIAL: NCT00091286
Title: Evaluation of the Immunogenicity of Vaccination With HER-2/Neu and CEA Derived Synthetic Peptides With GM-CSF-in-Adjuvant, in Patients With Stage IIB, III, or IV Colorectal Cancer
Brief Title: Vaccine Therapy in Treating Patients With Stage IIB, Stage III, or Stage IV Colorectal Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Slow accruals
Sponsor: Craig L Slingluff, Jr (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Craig L Slingluff, Jr, Director, Human Immune Therapy Center, University of Virginia
Organization: University of Virginia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9976; UVACC-GI37; UVACC-23302
Record Dates: First submitted 2004-09-07; First posted 2004-09-09 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage IIB colon cancer; stage IIIA colon cancer; stage IIIB colon cancer; stage IIIC colon cancer; stage IVA colon cancer; stage IVB colon cancer; recurrent rectal cancer; stage IIB rectal cancer; stage IIIA rectal cancer; stage IIIB rectal cancer; stage IIIC rectal cancer; stage IVA rectal cancer; stage IVB rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Receptor Protein-Tyrosine Kinases; Granulocyte-Macrophage Colony-Stimulating Factor

ARMS (1):
- Peptide Vaccine + Montanide + GM-CSF (Experimental): Colon peptide mixture (100 mcg each of the 4 peptides) plus 190 mcg of tetanus toxoid peptide, plus GM-CSF (110 mcg) in Montanide ISA-51 adjuvant
  Interventions: Biological: HER-2-neu, CEA peptides, GM-CSF, Montanide ISA-51 vaccine

INTERVENTIONS:
Biological: HER-2-neu, CEA peptides, GM-CSF, Montanide ISA-51 vaccine

SUMMARY:
RATIONALE: Vaccines made from peptides may make the body build an immune response to kill tumor cells.

PURPOSE: This clinical trial is studying how well vaccine therapy works in treating patients with stage IIB, stage III, or stage IV colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether vaccination comprising HER-2-neu and carcinoembryonic antigen synthetic peptides, sargramostim (GM-CSF), and Montanide ISA-51 causes an immune response in patients with stage IIB, III, or IV colorectal cancer.
* Determine the safety of this regimen in these patients.

OUTLINE: Patients receive vaccination comprising HER-2-neu and carcinoembryonic antigen synthetic peptides, sargramostim (GM-CSF), and Montanide ISA-51 on days 1, 8, and 15. On day 22, patients undergo removal of the lymph node into which the vaccination site drains to determine whether the immune system is responding to the vaccine.

PROJECTED ACCRUAL: A maximum of 15 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of colorectal cancer

  * Stage IIB, III, or IV disease
* HLA-A2- or -A3-positive

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,000/mm^3
* Hemoglobin > 9 g/dL
* Platelet count > 100,000/mm^3

Hepatic

* Liver function tests ≤ 2.5 times upper limit of normal (ULN)

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No New York Heart Association class III or IV heart disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known or suspected allergies to any component of the study drug
* No active connective tissue disease requiring medications
* No systemic autoimmune disease with visceral involvement
* No uncontrolled diabetes
* No other severe autoimmune disease
* No medical contraindication or potential problem that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 30 days since prior immunotherapy
* More than 30 days since prior growth factors
* More than 30 days since prior allergy shots
* No prior vaccination with any study peptides for malignancy

Chemotherapy

* More than 30 days since prior chemotherapy

Endocrine therapy

* More than 30 days since prior steroids

Radiotherapy

* More than 30 days since prior radiotherapy

Surgery

* More than 30 days since prior surgery

Other

* At least 30 days, but ≤ 24 months, since prior therapy for colorectal cancer
* No concurrent illegal drug use

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2003-03-24 (Actual); Primary Completion 2008-02-15 (Actual); Study Completion 2008-02-15 (Actual)

PRIMARY OUTCOMES:
Safety of the 4-peptide mixture | 30 days following last vaccine
  Adverse events
Number of patients with an immune response to the peptides | through Day 22
  T cell responses against the peptides as measured in the sentinel immunized node

SECONDARY OUTCOMES:
Immunogenicity of the peptide mixture measured in the peripheral blood | through Day 22
  T cell responses against the peptides and/or tumor

CONTACTS AND LOCATIONS:
Overall Officials: Charles M. Friel, MD, Study Chair — University of Virginia
Locations (1):
- University of Virginia Cancer Center, Charlottesville, Virginia, United States